CLINICAL TRIAL: NCT02482077
Title: Efficacy and Safety Study of Sofosbuvir Containing Regimens in Subjects With Chronic Hepatitis C Virus Genotype 2 Infection
Brief Title: Sofosbuvir Containing Regimens for the Treatment of Chronic HCV GT2 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_HCV G2 Study
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Sofosbuvir; Ribavirin; daclatasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SOF+RBV 8 wk (Experimental): Participants will receive SOF+RBV for 8 weeks.
  Interventions: Drug: SOF+RBV
- SOF+RBV 12 wk (Experimental): Participants will receive SOF+RBV for 12 weeks.
  Interventions: Drug: SOF+RBV
- SOF+DCV 8 wk (Experimental): Participants will receive SOF+DCV for 8 weeks.
  Interventions: Drug: SOF+DCV
- SOF+DCV 12 wk (Experimental): Participants will receive SOF+DCV for 12 weeks.
  Interventions: Drug: SOF+DCV
- LDV/SOF 8 wk (Experimental): Participants will receive LDV/SOF for 8 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF 12 wk (Experimental): Participants will receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: SOF+RBV — Sofosbuvir (SOF) 400 mg tablet administered orally once daily. Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg).
  Other Names: GS-7977; PSI-7977; Sovaldi®; Copegus®
  Arms: SOF+RBV 12 wk; SOF+RBV 8 wk
Drug: SOF+DCV — Sofosbuvir (SOF) 400 mg tablet administered orally once daily. Daclatasvir (DCV) 60mg tablet administered once daily.
  Other Names: GS-7977; PSI-7977; Sovaldi®; BMS-790052; Daklinza®
  Arms: SOF+DCV 12 wk; SOF+DCV 8 wk
Drug: LDV/SOF — Ledipasvir 90 mg /Sofosbuvir 400 mg (LDV/SOF) FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5885; Harvoni®
  Arms: LDV/SOF 12 wk; LDV/SOF 8 wk

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of Sofosbuvir containing regimens in treatment-naive or treatment-experienced patients with HCV genotypes 2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18 years, with chronic genotype 2 HCV infection;
2. Documented HCV treatment-naïve or treatment-experienced subjects who failed previous PEG+RBV regimen;
3. HCV RNA > 10,000 IU/mL at Screening;
4. Screening laboratory values within defined thresholds
5. Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

1. Pregnant or nursing female or male with pregnant female partner;
2. HIV or chronic hepatitis B virus (HBV) infection;
3. Hematologic or biochemical parameters at Screening outside the protocol-specified requirements;
4. Active or recent history (≤ 1 year) of drug or alcohol abuse;
5. Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks after discontinuation of therapy | Post treatment Week 12
  SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after last dose of study drug.
Proportion of participants with adverse events leading to permanent discontinuation of study drug(s) | Baseline up to Week 24

SECONDARY OUTCOMES:
Proportion of participants with unquantifiable HCV viral load at specified time points during and after treatment | Baseline up to Week 24
HCV RNA levels and change during and after treatment. | Baseline up to Week 24
Proportion of participants with on-treatment virologic breakthrough and relapse | Baseline up to Week 24
  Viral breakthrough is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment, but did not achieve a sustained virologic response (SVR). Viral relapse is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) within 4 weeks of end of treatment, but did not achieve an SVR.

CONTACTS AND LOCATIONS:
Overall Officials: George KK Lau, MD, Principal Investigator — Humanity and Health GI and Liver Centre
Locations (2):
- China (2):
  - Liver Fibrosis Diagnosis and Treatment Centre, 302 Hospital, Beijing, Beijing Municipality
  - Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong